CLINICAL TRIAL: NCT05203315
Title: A Multicenter, Single-Arm, Open-Label Study Evaluating the Safety, Tolerability, and Efficacy of Duobrii® Lotion in the Treatment of Mild Plaque Psoriasis in Adults
Brief Title: Investigator Initiated Trial to Study Duobrii® Lotion in the Treatment of Mild Plaque Psoriasis in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austin Institute for Clinical Research (Network)
Collaborators: OrthoDermatologics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDCR-000245
Record Dates: First submitted 2021-12-02; First posted 2022-01-24 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: Open Label Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group A (Experimental): Subjects whose baseline Itch and/or Burning/Stinging Score is less than 2 (moderate), one tube of Duobrii along with one jar of CeraVe cream, will be dispensed to the subject at the Baseline visit. The study participant will be instructed to apply the CeraVe cream to the treatment area twice daily and advised to apply a thin layer of the Duobrii only to the affected skin once daily in the evening.
  Interventions: Drug: Duobrii 0.01 % / 0.045 % Topical Lotion; Drug: CeraVe, Topical Cream
- Treatment Group B (Experimental): Subjects whose baseline Itch and/or Burning/Stinging Score is greater than or equal to 2 (moderate), in addition to one tube of Duobrii along with one jar of CeraVe cream, the participant will be given a tube of hydrocortisone 1% cream and instructed to apply to the treatment area twice daily for 5 days, along with CeraVe cream. Starting at day 6 and ongoing, subjects will be instructed to discontinue the hydrocortisone cream and initiate Duobrii application every night, while continuing the CeraVe cream twice daily.
  Interventions: Drug: Duobrii 0.01 % / 0.045 % Topical Lotion; Drug: CeraVe, Topical Cream

INTERVENTIONS:
Drug: Duobrii 0.01 % / 0.045 % Topical Lotion — Duobrii® lotion (halobetasol propionate [HP] and tazarotene [Taz] 0.01%/0.045%) is currently on the market for the treatment of moderate to severe stable plaque psoriasis, and is classified as a high potency (Class II) corticosteroid.
Drug: CeraVe, Topical Cream — CeraVe cream will be used twice daily (in the morning and again in the evening) by the study participant in conjunction with Duobrii and Hydrocortisone cream.

SUMMARY:
This study seeks to evaluate the safety, tolerability, and efficacy of topical Duobrii® Lotion in adult subjects with mild plaque psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a common disease of both males and females, that can range in severity from very mild to very severe. Patient age, severity of disease, and the type and extent of the body surface area are often taken into consideration when selecting therapy. There is not a cure for this particular disease and treatment options often focus on relieving moderate to severe symptoms associated with the disease.

Biologic treatments are often used to treat the symptoms of moderate to severe plaque psoriasis. These symptoms often include inflammation, induration, and scaling. However, this study aims to research Duobrii® Lotion for the treatment of mild stable plaque psoriasis in male and female adults.

Approximately 40 subjects who meet the study entry criteria will be enrolled. For those subjects whose baseline Itch and/or Burning/Stinging Score is <2 (moderate), one tube of Duobrii, along with one jar of CeraVe cream, will be dispensed to the subject at the Baseline visit. Both Duobrii and CeraVe cream will be applied topically to the affected areas (as determined by the investigator at baseline). Subjects will be advised to apply the CeraVe cream twice daily (in the morning, and again in the evening after applying Duobrii), and advised to apply a thin layer of Duobrii only to affected skin once daily in the evening.

For those subjects whose baseline Itch and/or Burning/Stinging Score is >=2 (moderate) in the treatment areas, in addition to being dispensed Duobrii and CeraVe, the participants will be given a tube of hydrocortisone 1% cream and instructed to apply to the treatment area twice daily for 5 days, along with CeraVe cream. Starting at day 6 and ongoing subjects will be instructed to discontinue the hydrocortisone cream and initiate Duobrii application every night, while continuing the CeraVe cream twice daily. Affected areas on the palms and soles, while not included in the Investigators Global Assessment, hereinafter referred to as IGA, or Body Surface Area, hereinafter referred to as BSA, assessment, are considered treatment areas and therefore are subject to the same guidelines for Itch and/or Burning/Stinging Scores as noted above.

Subjects will be instructed to make an unscheduled visit if the participant believes their psoriasis has cleared in between scheduled study visits, and will be allowed to discontinue the Duobrii if the investigator agrees their IGA=0 (clear). Subjects will be advised to restart Duobrii once the investigator determines the subject has an IGA=2 (mild). The duration of the study will be 28 weeks. The initial application will be made by the subject per instruction from the study staff either at the investigational center, or at their home. The subjects will be instructed to avoid exposure to direct sunlight, artificial ultraviolet light sources and to use protective clothing to prevent sunburn. Subjects will apply their once daily treatments at home as explained by the study coordinator or designee at each investigational center.

During post-baseline study visits (Weeks 2, 4, 6, 8, 12, 16, 20 and 24) the subjects will be asked to return their containers of Duobrii and CeraVe which will be evaluated for drug usage compliance. New containers will be dispensed as needed. During the study, subjects will be allowed to use investigator-approved non-medicated cleansers and sunscreens; no other skin care products will be permitted on the treatment areas. The investigator will assess the areas affected by psoriasis at each study visit.

All areas affected by psoriasis (excluding face, genitals, axillae, and intertriginous areas) are to be treated with Duobrii and CeraVe. Information on reported and observed adverse events (AEs) will be obtained at each visit.

For all female subjects of childbearing potential, urine pregnancy testing will be performed at Screening, Baseline, and each subsequent visit.

The Dermatology Life Quality Index questionnaire (DLQI) questionnaire will be administered to subjects at Day 0 (Baseline), each post-baseline visit, and the final visit. The DLQI will not be completed at the Screening visit, Phone contact visit, or Unscheduled visits.

Subjects who terminate study participation early will be asked to complete all Week 28 assessments, as appropriate, prior to commencement of any alternative therapy for psoriasis (if possible). Subjects who discontinue from the study during the treatment period will not be replaced and these subjects may be asked to return for the week 28 visit after the last treatment visit.

If signs or symptoms develop in the selected treatment areas during the treatment period that restrict daily activities or make continued application of Duobrii difficult due to discomfort, the investigator may instruct the subject to temporarily interrupt use of Duobrii and to resume application of Duobrii once the signs/symptoms have subsided. The investigator should try to minimize study drug interruptions; and if needed, make best efforts to limit a "drug holiday" to 5 days. If Duobrii interruption does exceed 5 consecutive days, the investigator may restart Duobrii at a decreased frequency. If Duobrii is interrupted, discontinued, or a concomitant medication is used to treat a sign/symptom, an adverse event shall be recorded.

Subjects who discontinue from the study due to AEs will return for the 28 week visit and will be instructed to follow-up with their primary care physician, if indicated. Any subject who has an AE during the treatment period will be followed by the investigator until resolution (return to normal or to the baseline state) or stabilization, as determined by the investigator.

In addition, application of study drug may be delayed or halted at any time if ongoing safety data evaluations (including reports of local skin reactions, such as skin atrophy, or severe AEs) raise concern for subject safety. If the subject participation is suspended, all the subject's safety data will be reviewed by the investigator to determine course of action.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of any race, at least 18 years of age.
2. Freely provides both verbal and written informed consent.
3. Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
4. Has a clinical diagnosis of stable plaque psoriasis at least 6 months before the Baseline visit, confirmed by prior medical documentation and/or according to the subject/caregiver report.
5. Has an IGA score of 2 at the Baseline visit. (The face, genitals, axillae, and intertriginous areas are to be excluded from this assessment, if psoriasis is present).
6. Is in good general health based on the subject's medical history.
7. If female and of childbearing potential, must have a negative urine pregnancy test at the Screening visit and Baseline visit prior to randomization.
8. IF female, is either not of childbearing potential, defined as postmenopausal for at least 12 months or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing 1 of the following methods of birth control throughout the study:

   * Condom with spermicide, diaphragm with spermicide, intrauterine device, or abstinence
   * Stable use of a hormonal contraceptive (oral, implant, insertable, injection or transdermal patch) for at least 3 months prior to the Baseline visit.
9. Subject is willing to comply with study instructions and return to the clinic for required visits.

Exclusion Criteria:

1. Has spontaneously improving or rapidly deteriorating plaque psoriasis or presence of guttate or pustular psoriasis, as determined by the investigator.
2. Presents with psoriasis that was treated with prescription medication and failed to respond to treatment, even partially or temporarily, as determined by the investigator.
3. Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator.
4. Is pregnant, nursing an infant, or planning a pregnancy during the study period.
5. Has received treatment with any investigational drug or device within 60 days or 5 drug half-lives (whichever is longer) prior to the Baseline visit, or is concurrently participating in another clinical study with an investigational drug or device. Subject may be enrolled in the follow-up phase of a COVID-19 vaccine trial.
6. Received treatment with any topical antipsoriatic drug product within 14 days prior to the Baseline visit.
7. Has used any phototherapy (including laser), photochemotherapy, or non-biologic systemic psoriasis therapy (such as newer oral psoriasis medications (eg Otezla), systemic corticosteroids, methotrexate, retinoids or cyclosporine) within 4 weeks prior to the Baseline visit.
8. Has used immunomodulatory therapy (biologics) known to affect psoriasis within 3 months of the Baseline visit.
9. Has had prolonged exposure to natural or artificial sources of ultraviolet radiation within 4 weeks prior to the Baseline visit or is intending to have exposure during the study thought likely by the investigator to modify the subject's psoriasis.
10. Is currently using lithium or Plaquenil.
11. Has a history of hypersensitivity or allergic reaction to any of Duobrii constituents.
12. Is unable to be compliant with study procedures, study drug administration requirements, study visit schedules, and prohibitions regarding the use of concomitant medications/therapies.
13. Is unable to communicate or cooperate with the investigator.
14. Has any underlying disease (e.g., uncontrolled diabetes, cardiac disease) that the investigator deems uncontrolled that poses a concern for the subject's safety while participating on the study.
15. Has a history of malignancy within 5 years before the Screening visit, except completely treated in situ carcinoma of the cervix or completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin with no evidence of recurrence in the past 12 weeks.
16. Has a planned or expected major surgical procedure during the clinical study.
17. Has a history of drug or alcohol abuse as determined by the investigator.
18. Is considered by the investigator, for any other reason, to be an unsuitable candidate for the study.
19. Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
20. Are employees of Bausch Health.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Treatment Success by Percent Investigators Global Assessment (IGA) | 28 Weeks
  The primary efficacy endpoint will be the percent of subjects with treatment success, defined as an Investigators Global Assessment (IGA) score equating to "Clear". 0: Clear, 1: Mild, 2: Moderate, 3: Severe.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, MBA, Principal Investigator — Austin Institute for Clinical Research; Megan Couvillion, MD, Principal Investigator — Austin Institute for Clinical Research
Locations (2):
- United States (2):
  - Austin Institute for Clinical Research, Inc., Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas